CLINICAL TRIAL: NCT02767102
Title: Serum and Salivary Melatonin Levels and Antioxidant Power of Melatonin-rich Red Wine
Brief Title: Bioavailability and Bioactivity of Red Wine Melatonin in Humans
Acronym: Wine-MLT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Milan (Other)
Responsible Party: Principal Investigator, ANDREA SARDELLA, Associate Professor, University of Milan
Allocation: Randomized | Model: Crossover | Masking: Quadruple
Other Study IDs: Red Wine Melatonin
Record Dates: First submitted 2016-04-30; First posted 2016-05-10 (Estimated); Last update posted 2016-05-10 (Estimated); Status verified 2016-05

CONDITIONS: Bioavailability
Keywords: Mediterranean diet; indoleamine; nutraceuticals; nutrition; oxidative stress
MeSH Terms: interventions — Melatonin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Red wine with Melatonin (Experimental): Rosso di Marco is a wine without MLT (previous screening). This wine will be enriched with 10 ng mL-1 MLT (MLT+) and used as experimental wine.
  Interventions: Other: Red wine with melatonin
- Red wine without Melatonin (Placebo Comparator): Rosso di Marco is a wine without MLT (previous screening). This wine will be used as placebo treatment (PLC).
  Interventions: Other: Red wine without melatonin

INTERVENTIONS:
Other: Red wine with melatonin — Twelve healthy volunteers will be recruited to receive both 125 mL of red wine rich in MLT (10 ng mL-1)
  Arms: Red wine with Melatonin
Other: Red wine without melatonin — Twelve healthy volunteers will be recruited to receive both 125 mL of red wine without MLT
  Arms: Red wine without Melatonin

SUMMARY:
Melatonin (MLT) is a bioactive compound in red wine. The investigators will investigate the serum and salivary concentrations and antioxidant power of MLT after the intake of a glass of red wine. Twelve healthy volunteers were recruited to receive both 125 mL of red wine rich in MLT (10 ng mL-1) and without MLT (placebo), via a randomized, cross-over, and double-blind design. Serum and salivary MLT will be measured by liquid chromatography coupled to mass spectrometry (LC-MS) and enzyme-linked immunosorbent (ELISA), respectively. The ferric ion reducing antioxidant power (FRAP) will be analyzed.

DETAILED DESCRIPTION:
Melatonin (MLT) is a bioactive compound in red wine. No information is currently available on serum and salivary concentrations of MLT after drinking a glass of red wine, containing this indoleamine. Hence, in this study, the investigators will investigate the levels of MLT, in serum and saliva, soon after the intake of the MLT-rich red wine, and, correspondingly, they will verify the antioxidant power of the same biological fluids.

This will be a randomized, crossover, double-blind, placebo-controlled study with two treatment arms. Twelve healthy volunteers will be recruited to receive both 125 mL of red wine rich in MLT (10 ng mL-1) and without MLT (placebo), via a randomized, cross-over, and double-blind design.

Serum and salivary MLT will be measured by liquid chromatography coupled to mass spectrometry (LC-MS) and enzyme-linked immunosorbent (ELISA), respectively. The ferric ion reducing antioxidant power (FRAP) will be also analyzed.

For serum analyses, samples will be collected at 0, 30, 60 and 90 min. For saliva analyses, samples will be collected at 0, 45 and 120 min.

ELIGIBILITY:
Inclusion Criteria:

* to be healthy
* to have normal weight (BMI 18.5-25.0)
* to voluntarily accept to participate to the study.

Exclusion Criteria:

* pregnancy and lactation for women;
* supplementation with MLT and/or any other dietary supplement (vitamins, antioxidants, botanicals, phytochemicals)
* systemic and chronic-degenerative diseases
* abnormal hematological parameters
* heavy smoking and alcohol drinking
* high-intensity physical activity
* under pharmacological treatment

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2014-07; Primary Completion 2015-03 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Serum and salivary melatonin after red wine intake (with or without MLT) | Time-course of the serum melatonin levels in healthy volunteer from 0 min to 90 min after administration of red wine. Time-course of the salivary melatonin levels in healthy volunteer from 0 min to 120 min after administration of red wine.
  LC-MS analyses for serum and ELISA analyses for saliva

SECONDARY OUTCOMES:
Antioxidant power of saliva and serum after red wine intake (with or without MLT) | Time-course of the serum antioxidant power in healthy volunteer from 0 min to 90 min after administration of red wine. Time-course of the salivary antioxidant power in healthy volunteer from 0 min to 120 min after administration of red wine.
  FRAP analyses

OTHER OUTCOMES:
Adverse effects | Acute side effects during the trial recorded at each experimental day each experimental day, up to 1 day after
  Questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- University of Milan, Milan, Italy, Italy

IPD SHARING:
Plan to Share IPD: No